CLINICAL TRIAL: NCT05223140
Title: Optimal Time Intervals for Vaginal Breech Births: A Multi-Site Case-Control Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 309591
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Intensive Care, Neonatal; Perinatal Death
Keywords: Physiological Breech Birth Algorithm; premature cord clamping; NICU; early perinatal death
MeSH Terms: conditions — Perinatal Death | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Admission to NICU or early perinatal death
  Interventions: Behavioral: Birth within 7 minutes of rumping; Behavioral: Premature cord clamping
- Controls: No admission to NICU or early perinatal death
  Interventions: Behavioral: Birth within 7 minutes of rumping; Behavioral: Premature cord clamping

INTERVENTIONS:
Behavioral: Birth within 7 minutes of rumping — Birth within 7 minutes of rumping (+3 station), within 5 minutes of birth of pelvis, within 3 minutes of birth of umbilicus
  Other Names: Adherence to physiological breech birth algorithm
Behavioral: Premature cord clamping — Umbilical cord clamping <1 minute following birth
  Other Names: Immediate cord clamping

SUMMARY:
This study uses a case-control design to test the hypotheses that avoidable delay in late second stage and premature cord clamping are associated with admission to the neonatal unit and/or early perinatal death following vaginal breech births. We aim to determine the predictive value of: 1) adherence/non-adherence to the Physiological Breech Birth Algorithm; and 2) premature cord clamping (<1 minute following birth) for admission to the neonatal unit and/or perinatal death following vaginal breech births. The secondary objectives are to: 1) test all variables for a single-factor association with the primary outcome; and 2) test the predictive values of associated variables using linear regression; in order to 3) explore other factors contributing to adverse outcomes in vaginal breech births.

DETAILED DESCRIPTION:
This study replicates a previous successful pilot study (Spillane et al 2021). The sample size calculation for the original study was based on the hypothesis that among those breech births where a neonatal death or admission to the neonatal intensive care unit (NICU) occurs following the birth, the time between the birth of the fetal pelvis and the birth of the aftercoming head will be greater than three minutes more often than it is among the controls, where no death or NICU admission has occurred. The hypothesis was developed from what is already known from previous research by Reitter, Halliday and Walker (2020). The study found that the time between the birth of the pelvis and the birth of the aftercoming head is more than three minutes in only 25% per cent of breech births with good outcomes. Spillane et al's study hypothesised that this interval would be more than three minutes in 75% of births where death or a NICU admission occurred.

Spillane et al's power calculation determined that a sample size of fifteen cases and thirty controls would be required to infer an association between a pelvis to head interval of >3 minutes and the composite neonatal outcome (death or NICU admission), with a confidence interval of 95% and a power of 80%. The results of that study confirmed that association (p=<.0005).

We have not re-calculated sample size. Our aims in this study are to confirm the results of the original study by replication in multiple different settings and to explore additional confounding variables that may only be apparent in larger data sets. We are particularly interested in the influence of immediate cord clamping on these outcomes, but it was not possible to calculate a sample size based on the original study due to none of the cases having anything other than immediate cord clamping (n=0). Therefore, we are seeking a larger sample size in the hopes of being able to identify an appropriate sample size for future research, and to confirm the results of the previous study.

All anonymised data gathered in each site will be combined and analysed as a single data set by the Co-Investigators. The complete anonymised data set, combining data from all sites, will be downloaded and stored within the KCL Sharepoint for analysis.

We will first calculate the time to event interval for all variables of interest and report descriptive statistics for all variables, including means, medians and range for continuous variables. Exposures and confounders will also be converted into binary variables, reflecting the cut-offs used in the Physiological Breech Birth Algorithm. These will then be tested against the primary outcome using the non-parametric chi-square, or Fisher's Exact tests where cell frequencies are too small for the chi-square test.

Linear and logistic regression analysis will be used to test the predictive values of meeting or exceeding the recommended time limits in the Physiological Breech Birth Algorithm, and of maintaining and intact umbilical cord until the onset of respiration or not. Further linear and logistic regression analyses will be conducted with all variables that show an association with the composite neonatal outcome to determine their predictive value, and additional variables to explore their potential as confounding factors for investigation in future studies.

ELIGIBILITY:
CASES

INCLUSION CRITERIA:

* Singleton pregnancy > 37+0 weeks with a breech-presenting fetus born vaginally;
* Alive on admission to intrapartum care
* Admission to the neonatal unit or early neonatal death (within 6 days of birth);
* Healthcare professional in attendance.

EXCLUSION CRITERIA

* Births which took place prior to the arrival of a trained health care professional;
* Major congenital anomaly, identified prior to or after birth, likely to have compromised neonatal condition.

CONTROLS

INCLUSION CRITERIA:

* Singleton pregnancy > 37+0 weeks with a longitudinal breech-presenting fetus born vaginally;
* No admission to the neonatal unit or early neonatal death (within 6 days of birth);
* Healthcare professional in attendance;
* Occurring immediately prior to the matched case; and
* Matched for parity with that case (nullip/multip).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Vaginal breech births will be identified by the local PI, who is a member of the clinical care team, through a search of routine electronic healthcare records. Once vaginal breech births have been identified, the primary outcome will be identified for each record in time-descending order, beginning with the most recent vaginal breech birth. When a case (NICU admission or neonatal death) is identified, then two controls will be identified in time-descending order and matched for parity with the case. Only the medical records which have been identified as cases and controls for the study will be accessed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Admission to neonatal unit | Immediately following a vaginal breech birth
  Admission to intensive care or special care neonatal unit
Early perinatal death | Within 6 days following a vaginal breech birth
  Neonatal death
Composite primary outcome | Up to 6 days following birth
  Neonatal death or admission

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Walker, Principal Investigator — King's College London
Locations (5):
- United Kingdom (5):
  - Chelsea and Westminster Hospital, London
  - West Middlesex Hospital, London
  - Frimley Health NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Kingston University Hospital NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data will also be uploaded onto an online open access repository as part of the publication process, to ensure sufficient peer review and public scrutiny. Published results will not contain any personal data that could allow identification of individual participants or the location of the births included in the analysis.
Supporting Information: Study Protocol, CSR
Time Frame: Study Protocol -- on registration Clinical Study Report -- on publication
Access Criteria: Data will be available for 10 years